CLINICAL TRIAL: NCT03753685
Title: Efficacy and Safety of X-396(Ensartinib) in ALK-Positive NSCLC Patients With Brain Metastases: A Phase Ⅱ, Open-Label, Single Arm, Multicenter Study
Brief Title: X-396(Ensartinib) Capsules in ALK-Positive NSCLC Patients With Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chang Jian Hua, Director, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTP-42324-IIT
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Nonsmall Cell Lung Cancer; Brain Metastases
Keywords: NSCLC; Brain metastases; ALK mutations; X-396 (Ensartinib)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Capsules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- X-396(Ensartinib) Capsule (Experimental)
  Interventions: Drug: X-396(Ensartinib) Capsule

INTERVENTIONS:
Drug: X-396(Ensartinib) Capsule — All consented, enrolled, eligible patients receive X-396 capsules, 225mg once daily.

SUMMARY:
To assess efficacy and safety of oral X-396 (Ensartinib) capsule in Chinese ALK-positive NSCLC patients with brain metastases, eligible patients will be enrolled with objective responses being primary outcome measures.

DETAILED DESCRIPTION:
In this phase Ⅱ, open-label, single arm, multicenter study, efficacy and safety of oral X-396 capsule (Ensartinib) in 37 Chinese ALK-positive NSCLC patients with brain metastases will be assessed. Eligible patients will receive 225mg X-396 capsules once daily and objective responses of brain metastasis based on investigator assessment according to Response Assessment in Neuro-Oncology (RANO) are primary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed locally advance or recurrent/metastatic NSCLC that was positive for ALK mutations.

  2. Contrast-enhanced MRI or CT confirmed parenchymal brain metastases with at least one measurable lesion (according to RANO and RECIST 1.1), which was not previously treated with radiotherapy.

  3. At most once treated with chemotherapy, which must have been completed at least 4 weeks before the initiation of study treatment. Any adverse events related to previous chemotherapy treatment have disappeared.

  4. Female or male, 18 years of age or older 5. A Karnofsky Performance Status score of at least 60. 6. An expected survival time of at least 12 weeks. 7. Adequate organ functions, defined as absolute neutrophils count ≥1.5*10^9/L，platelets count ≥80*10^9/L, hemoglobin concentration≥ 9 g/dL, total bilirubin ≤1.5 *ULN (upper limits of normal), ALT≤2.5 *ULN, AST≤2.5 *ULN, creatinine≤1.5 *ULN.

  8. Drug related toxicities has been relieved to grade 1 (based on NCI CTCAE v4.03), except for hair loss.

  9. Being willing and able to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

  10. Signed and dated informed consent.

Exclusion Criteria:

* 1. Currently under treatment of other systemic anti-cancer therapies. 2. Evidence of active malignancy within last 5 years. 3. Patients who participated in other clinical trials within last 4 weeks before the initiation of study treatment.

  4. Patients who received surgery or immunotherapy within last 4 weeks before the initiation of study treatment, or received radiotherapy within last 2 weeks before the initiation of study treatment.

  5. Patients who previously received organ transplantation or stem cell transplantation.

  6. Patients with clinically significant cardiovascular and cerebrovascular diseases.

  7. Patients with dysphagia, active gastrointestinal diseases or other conditions that will interfere significantly with the absorption, distribution, metabolism or excretion of study medication.

  8. Patients who are active carrier of hepatitis B (HBsAg positive and HBV-DNA ≥500IU/mL), hepatitis C virus antibody, treponema pallidum antibody or HIV antibody.

  9. Patients with interstitial lung disease history or signs of active interstitial lung disease.

  10. Pregnant and lactating women. 11. Patients with known allergy or delayed hypersensitivity reaction to study drug or its excipients.

  12. Patients who need to receive drugs which could induce QT/QTc interval prolongation or torsade de pointes, or drugs which are potent CYP3A4 inhibitors or inducers within last 14 days before the initiation of study treatment and during the study.

  13. Patients who are currently under treatment of warfarin or other coumarin anticoagulants.

  14. Patients with other illness or medical conditions potentially interfering with the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial objective response rate (iORR) based on investigator assessment according to RNAO-BM. | 12 weeks
  iORR per RANO-BM calculated as the proportion of patients with a best intracranial overall response defined as complete response (CR) or partial response (PR), based on investigator assessment.

SECONDARY OUTCOMES:
Disease control rate based on intracranial response (iDCR) according to RANO-BM. | 12 weeks
  Defined as the percentage of patients who have achieved intracranial overall response of CR, PR and stable disease (SD), assessed by investigator.
Progression-free survival based on intracranial response (iPFS) according to RANO-BM | 36 months
  Defined as time from first dose of X-396 capsule to intracranial disease progression or death due to any causes, assessed by investigator.
Time to progression based on intracranial response (iTTP) according to RANO-BM. | 36 months
  Defined as time from first dose of X-396 capsule to intracranial disease progression, assessed by investigator.
Duration of response based on intracranial response (iDOR) according to RANO-BM. | 36 months
  Defined as time from documentation of intracranial response (CR or PR) to intracranial disease progression or death, assessed by investigator.
Intracranial objective response rate (iORR) based on intracranial response according to RECIST 1.1 | 12 weeks
  iORR per RECIST 1.1 calculated as the proportion of patients with a best intracranial overall response defined as complete response (CR) or partial response (PR), based on investigator assessment.
Disease control rate based on intracranial response (iDCR) according to RECIST 1.1 | 12 weeks
  Defined as the percentage of patients who have achieved intracranial overall response of CR, PR and stable disease (SD), assessed by investigator.
Progression-free survival based on intracranial response (iPFS) according to RECIST 1.1 | 36 months
  Defined as time from first dose of X-396 capsule to intracranial disease progression or death due to any causes, assessed by investigator.
Time to progression based on intracranial response (iTTP) according to RECIST 1.1 | 36 months
  Defined as time from first dose of X-396 capsule to intracranial disease progression, assessed by investigator.
Duration of response based on intracranial response (iDOR) according to RECIST 1.1 | 36 months
  Defined as time from documentation of intracranial response (CR or PR) to intracranial disease progression or death, assessed by investigator.
Objective response rate (ORR) based on overall response according to RECIST 1.1. | 12 weeks
  ORR per RECIST 1.1 calculated as the proportion of patients with a best overall response defined as complete response (CR) or partial response (PR), based on investigator assessment.
Disease control rate based on overall response (DCR) according to RECIST 1.1 | 12 weeks
  Defined as the percentage of patients who have achieved overall response of CR, PR and stable disease (SD), assessed by investigator.
Progression-free survival based on overall response (PFS) according to RECIST 1.1 | 36 months
  Defined as time from first dose of X-396 capsule to overall disease progression or death due to any causes, assessed by investigator.
Time to progression based on overall response (TTP) according to RECIST 1.1 | 36 months
  Defined as time from first dose of X-396 capsule to overall disease progression, assessed by investigator.
Duration of response based on overall response (DOR) according to RECIST 1.1 | 36 months
  Defined as time from documentation of overall response (CR or PR) to overall disease progression or death, assessed by investigator.
Overall survival (OS) | 36 months
  Defined as time from first dose of X-396 to death due to any causes.
Incidence of patients experiencing adverse events. | 36 months
  Incidence of adverse events occurred during the study (from the timeoint of signing a informed consent form to 30days after the end of trial).

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy Of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No